CLINICAL TRIAL: NCT00752037
Title: Safety and Efficacy of Lopinavir/Ritonavir in Combination With Raltegravir in HIV-infected Patients
Brief Title: Safety Study of Lopinavir/Ritonavir With Raltegravir in HIV-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Michael's Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: JIhad Slim,Md, Saint Michael's Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INV 08/08
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: HIV; Protease Inhibitor; Integrase Inhibitor; Treatment Experienced; Naive
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir; Raltegravir Potassium; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): open label single arm
  Interventions: Drug: lopinavir/ritonavir and raltegravir

INTERVENTIONS:
Drug: lopinavir/ritonavir and raltegravir — lopinavir/ritonavir 400/100 mg po b.id. in combination with raltegravir 400 mg po b.i.d.
  Other Names: Kaletra, Isentress

SUMMARY:
A single center, open label, 48-week study of lopinavir/ritonavir in combination with raltegravir. 30 patients, both naïve and experienced, will be enrolled. 15 treatment naïve patients and 15 treatment experienced patients enrolled

DETAILED DESCRIPTION:
This is an open-labeled, non-randomized exploratory trial in selected volunteers who meet the stated enrollment criteria. This study will assess the impact of lopinavir/ritonavir in combination with raltegravir on HIV-1

Patients will be evaluated frequently over the 52 weeks of the protocol. Patients will be seen at screening, baseline, week 4, 12, 24, 36, 48, and 52, to include physical examination, assessment for the development of AIDS-defining conditions, hematology, chemistry, lipid profile, CD4, CD8 cell counts, plasma HIV-1 RNA ultrasensitive, and assessment of adverse events. If HIV-1 RNA becomes detectable, this will be repeated for confirmation with 2 weeks. HIV genotyping and phenotyping will be performed on patients who demonstrate repetitive plasma viral load levels of > 1,000 copies/mL.

An interim analysis will be performed when all patients have reached the week 24 visit.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit, and confirmed by Western blot, positive HIV-1 blood culture, positive HIV serum antigen, or plasma viremia at any time prior to study entry. If no record exists, testing must occur at screening.
2. Males and non-pregnant females > 18 years of age. (Children are being excluded as they are immunologically different than adults)
3. HIV-1 RNA > 1000 copies/ml for both patient naive and experienced to antiretroviral therapy in order for phenotypic susceptibility to be performed. There in no inclusion criteria for CD4 count.
4. Treatment experienced patients , defined as having taken medications from two of the following three classes of antiretrovirals: NRTI, NNRTI, or PI must have phenotypic susceptability to lopinavir/ritonavir as resulted by Phenosense GT
5. Laboratory tests ( Cbc w/diff, comprehensive metabolic panel) within pre-specified limits
6. Able to sign the informed consent, and is willing to comply with the requirements of this clinical trial.
7. Available for at least 52 weeks of follow up
8. If female and of child bearing potential must consent to remain abstinent throughout the study period and for 30 days after the last dose of study medications.( this is standard language)

Exclusion Criteria:

1. Pregnant or breast-feeding woman (pregnant women are being excluded as drug kinetics are different in pregnancy and the dynamics of immune reconstitution are unknown in this group)
2. Current treatment for malignancy other than basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or isolated cutaneous Kaposi's Sarcoma that is not being treated; those with prior cancer diagnosis, such as lymphomas must have been disease-free for at least 5 years
3. Absolute neutrophil count < 500, platelet count < 50,000, hemoglobin < 8 gm/dL
4. Evidence of end-organ disease, defined as follows: renal (calculated creatinine clearance of less than 50 mL/min); liver (liver-associated enzymes > 3 times the upper limits of normal)
5. Grade 3 (ACTG Grading Scale) or higher cholesterol or triglyceride elevations
6. Acute, serious infection requiring prescription drug therapy within 30 days prior to study entry
7. In the opinion of the investigator, there is evidence of an active ongoing opportunistic infection
8. Must not currently be undergoing treatment for an opportunistic infection.
9. Use of immune stimulation agents known to impact CD4 cell count in the peripheral circulation, to include IL2, interferon, G-CSF, GM-CSF, etc.
10. Use of immune suppressant drugs, with the exception of < 10 mg/day of prednisone .
11. Unwillingness to remain abstinent for duration of study
12. Experimental vaccines, to include HIV vaccines.
13. Patient who is currently enrolled in an experimental protocol, or is receiving an experimental medication.
14. Patients on 2 NRTIs with an NNRTI and a PI combination will not be allowed in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to evaluate the percentage of patients with HIV-1 RNA below 50 copies at week 48 receiving lopinavir/ritonavir in combination with raltegravir | week 48

SECONDARY OUTCOMES:
To evaluate the effect of lopinavir/ritonavir in combination with raltegravir in maintaining virological suppression | weeks 12, 24, 36, and 48
To evaluate the change from baseline in plasma HIV-1 RNA at weeks 12, 24, 36, and 48 | weeks 12, 24, 36, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Slim, MD, Principal Investigator — Saint Michael's Medical Center
Locations (1):
- Saint Michael's Medical Center, Newark, New Jersey, United States